CLINICAL TRIAL: NCT01650649
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple Ascending Dose Study to Assess the Safety, Tolerability, and Electrocardiographic Effects of Lofexidine When Administered Orally to Methadone Maintained Adult Subjects
Brief Title: Main Study of Lofexidine and Methadone Pharmacodynamic Interaction in Methadone Maintained Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: USWM, LLC (dba US WorldMeds) (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: USWM-LX1-1005-2; 1U01DA030916-01 (NIH)
Record Dates: First submitted 2012-07-09; First posted 2012-07-26 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Opioid Dependence; Methadone Withdrawal Syndrome
Keywords: lofexidine; methadone; interaction; pharmacodynamic; ECG; QTc
MeSH Terms: conditions — Opioid-Related Disorders | interventions — lofexidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lofexidine Titration in Methadone Maintained Subjects (Active Comparator): Methadone maintained subjects will be titrated on lofexidine up to the target therapeutic dose of 0.8 mg QID (4 tablets QID) or to the highest level tolerated. Following this initial titration attempt, all subjects will have their methadone dose reduced by 50% and lofexidine titration efforts will resume.
  Interventions: Drug: Lofexidine HCl
- Placebo titration in methadone maintained subjects (Placebo Comparator): Methadone maintained subjects will be titrated on placebo tablets in ascending doses of 1 tablet starting with 2 tablets (e.g. Day 1 2 tablets QID, Day 2 3 tablets QID, etc) to mimic titration for subjects randomized to lofexidine.
  Interventions: Drug: Lofexidine-matching sugar pill

INTERVENTIONS:
Drug: Lofexidine HCl — Lofexidine HCl 0.2 mg tablets titrated in ascending doses of 0.2 mg (1 tablet) QID starting at 0.4 mg (2 tablets) QID [e.g. Day 1 0.4 mg (2 tablets) QID, Day 2 0.6 (3 tablets)QID, etc] as described in the treatment arm. Option to down-titrate to 0.2 mg (1 tablet) QID if 0.4 mg (2 tablets) QID dose not initially tolerated.
  Arms: Lofexidine Titration in Methadone Maintained Subjects
Drug: Lofexidine-matching sugar pill — Lofexidine-matching sugar pill tablets titrated in ascending doses of 1 tablet starting at 2 tablets QID (e.g. Day 1 2 tablets QID, Day 2 3 tablets QID, etc)as described in the treatment arm. Option to down-titrate to 1 tablet QID if 2 tablets not initially tolerated.
  Arms: Placebo titration in methadone maintained subjects

SUMMARY:
The primary objective of this study is to assess QTc (an interval of the heart rhythm) interaction effects between lofexidine and methadone. The secondary objectives of the study are to evaluate the safety and tolerability of lofexidine by evaluating and monitoring pharmacokinetics (amounts of drug in the blood), vital signs (heart rate and blood pressure) and adverse events (side effects) when co-administered with methadone; to describe effects on opiate withdrawal when lofexidine is introduced following a 50% methadone dose reduction, as required to elicit a withdrawal response; and to evaluate the QTc interaction effects of lofexidine compared with placebo. The investigators hypothesize that while both agents (lofexidine and methadone) are known to prolong the QTc interval, the combination of the drugs will not create an additive effect which creates a significant safety concern. The investigators further hypothesize that subjects will be able to tolerate the therapeutic dose of lofexidine (0.8 mg four times daily) when the methadone maintenance dose is lowered to elicit withdrawal.

DETAILED DESCRIPTION:
This will be a randomized, double-blind, placebo-controlled multiple ascending dose study to assess the safety, tolerability, and electrocardiographic effects of lofexidine in 24 methadone-maintained adult subjects. The study will include a Screening Visit, an Inpatient Treatment Visit, and a Follow-Up Visit. Subjects will be randomized in 3:1 ratio to receive up to 4 tablets of lofexidine (0.2 mg/tablet) QID or 4 tablets matching placebo QID.

Subjects who are on a stable dose of methadone (80 - 120 mg/day) and who satisfy inclusion and exclusion criteria will be eligible for the study. Within 21 days of the Screening Visit, subjects will report to the inpatient study facility to begin the Inpatient Treatment Visit which will last between approximately 11 to 21 days. This visit will include an inpatient check-in (1 day), Methadone Baseline (1 day), Initial Lofexidine Titration (3 to 5 days), 1 or 2 Lofexidine Plateaus (2 to 4 days), Methadone Reduction (2 to 6 days) and Methadone Re-Titration and Discharge (2 to 4 days). The order of steps subjects will proceed through during the Inpatient Treatment Visit will vary depending on whether subjects are able to titrate to the highest dose of lofexidine or placebo during the Initial Lofexidine Titration. The highest dose of lofexidine (or placebo) will be 4 tablets QID (0.2 mg lofexidine per tablet or placebo) for a total daily lofexidine dose of 16 tablets (3.2 mg or placebo). Diagrams for the two scenarios that can occur with lofexidine titration are located in Figure 1 and 2 in the body of the protocol.

During the Methadone Baseline phase subjects will take a single daily dose of methadone at 1 PM and undergo baseline study assessments including electrocardiogram (ECG) monitoring, blood collection for methadone pharmacokinetics, and opiate withdrawal assessments (Clinical Opiate Withdrawal Scale, COWS and Short Opiate Withdrawal Scale, SOWS). The next day subjects will proceed to the Initial Lofexidine Titration phase. Subjects will continue using their baseline methadone dose. Lofexidine will be initiated at 2 tablets (0.4 mg or placebo) QID and titrated in daily increments of a single tablet (0.2 mg or placebo) QID to a total daily dose of 0.8 mg QID (or placebo), if tolerated by the subject. Lofexidine doses will escalate daily unless at any point the subject meets protocol-defined dose hold criteria (described below), which will trigger a reduction in dose to the previous highest tolerated dose (or to the 1 tablet dose, 0.2 mg or placebo, if subjects cannot tolerate the initial 2 tablets). Once subjects have titrated to the highest dose (ie, 4 tablets QID) or once the highest tolerated dose has been determined, they will proceed to a 2-day Lofexidine Plateau phase during which they will continue to receive their methadone maintenance dose. If the subject is unable to titrate up to 4 tablets QID (0.8 mg or placebo), the subject will continue to receive their highest tolerated dose in equal increments (eg, 2 or 3 tablets QID at 8AM, 1PM, 6PM, 11PM) for both days of the plateau. If the subject tolerates 4 tablets QID (0.8 mg or placebo), on the first day they will receive the 4 tablets QID (0.8 mg or placebo) according to the normal dosing schedule. On the second day, the lofexidine dosing schedule will be modified with subjects receiving a 1 tablet (ie, 0.2 mg or placebo) increase of the 1 PM lofexidine dose (5 tablets: 1 mg or placebo) and a 1 tablet (0.2 mg or placebo) reduction in the subsequent lofexidine dose (3 tablets: 0.6 mg or placebo) with the other 2 doses of 4 tablets (0.8 mg or placebo) for a total daily dose of 16 tablets (3.2 mg/day or placebo). On the second day of the Lofexidine Plateau phase, subjects will undergo electrocardiogram (ECG) monitoring and blood collection for methadone and lofexidine pharmacokinetics. COWS and SOWS assessments will be performed on both days of the Lofexidine Plateau.

Subjects who are titrated to a daily dose of 4 tablets (0.8 mg or placebo) QID while receiving their full dose of methadone will undergo a 4-day methadone dose reduction of 50% while continuing to take lofexidine or placebo at a daily dose of 16 tablets to evaluate the effects of lofexidine on methadone withdrawal signs and symptoms. These subjects who complete the initial Lofexidine Plateau at a dose of 0.8 mg lofexidine (or placebo) QID and who reach a COWS of 5 or greater prior to the fourth day of the reduced methadone dose administration may proceed early to Methadone Re-titration and Discharge at the Investigator's discretion. If the COWS score does not reach 5 within 4 days, the subject will proceed to Methadone Re-titration and Discharge.

Subjects who are unable to titrate to the highest lofexidine dose (4 tablets: 0.8 mg or placebo QID) while receiving their full dose of methadone will undergo a methadone dose reduction of 50% for up to 6 days while continuing to receive their highest tolerated dose of lofexidine from the initial titration. On the fourth day (or earlier at the investigator's discretion based on withdrawal response), lofexidine titration will resume by adding an incremental 1 tablet (0.2 mg or placebo) QID to the previously established tolerated dose up to the maximum 4 tablet (0.8 mg or placebo) QID dose. During these subsequent titration attempts lofexidine (or placebo) doses will escalate daily beginning on the fourth day of the reduction (or earlier based on discretion of the investigator) unless in any event a subject meets protocol defined dose-hold criteria (described below), which will trigger a reduction in dose to the previous highest tolerated dose and will require the Lofexidine Plateau procedures described above to be repeated while maintaining the subject on their newly reduced methadone dose (eg, 50% of their maintenance dose). Subjects who are unable to titrate to a higher lofexidine dose during the 50% Methadone Reduction than the dose they titrated to during the Initial Lofexidine Titration will not repeat the Lofexidine Plateau procedures.

During Methadone Reduction (whether for subjects entering an experimental 4-day 50% withdrawal phase at the tolerated 4 tablet [0.8 mg or placebo] QID lofexidine dose or for subjects continuing lofexidine titration at 50% methadone reduction), COWS and SOWS assessments of opiate withdrawal will be performed.

Following completion of the Lofexidine Plateau (repeated as necessary) and Methadone Reduction, subjects will begin the Methadone Re-Titration and Discharge phase during which lofexidine or placebo will be discontinued and methadone will be re-titrated to the starting dose (or to a higher or lower dose relative to baseline as medically indicated at the discretion of the investigator). Lofexidine may be used to treat withdrawal symptoms, if necessary. Following successful methadone titration and completion of study assessments, subjects will be discharged from the inpatient study clinic.

Subjects will return to the study clinic for a follow-up visit 7 days (±2 days) following clinic discharge for safety follow-up and adverse event collection. Subjects will be discharged from the study at this time unless they are medically unstable on their dose of methadone. Subject may be medically followed at a regular interval, as determined by the investigator, until the subject is considered sufficiently stable for study discharge.

Subjects who withdraw consent or meet any one of the following study termination criteria prior to completion of the study will be withdrawn. Study termination criteria will apply only to pre-dose readings. Baseline values for vital signs and ECG readings refer to values obtained at the time subjects are admitted to the clinic.

1. Cardiovascular events including the following:

   1. Systolic blood pressure (SBP) <70 mmHg and >20% below baseline value (if subject is asymptomatic, SBP termination criteria <70 mmHg)*
   2. Diastolic blood pressure (DBP) <40 mmHg and >20% below baseline value (if subject is asymptomatic, DBP termination criteria <30 mmHg)*
   3. Heart rate (HR) <40 bpm and >20% below baseline value (if subject is asymptomatic, HR termination criteria <30 bpm)*
   4. QTc >500 msec or >25% above baseline value for both males and females*
   5. Absolute QTcF>500 ms in females or >480 ms in males with a concurrent increase in average QTcF value >60 ms from the baseline value
   6. Persistent increase in QTcF >60 ms above baseline or persistent QTcF≥480 ms and ≤500 ms and electrolytes are normal
   7. Absolute QRS>120 ms along with a 25% increase from baseline
   8. Absolute PR>240 ms along with a 25% increase from baseline
   9. Syncope
   10. Clinically significant arrhythmia (including telemetry indication of ventricular tachycardia, ventricular fibrillation, Torsade de Pointes, 2nd degree AV block)* *ECGs and vital signs may be repeated as appropriate to confirm values and rule out extraneous results.
2. Serious medical problems thought to be related or unrelated to the study medications.
3. Intercurrent illness or medical complications that, in the opinion of the site investigator, preclude safe administration of study medications.

At the time of termination from the study, subjects will be discontinued from lofexidine or placebo; however, they may remain inpatient for up to 4 days while their methadone maintenance dose is re-titrated to their pre-study maintenance dose.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male and/or female, 18 to 60 years of age (inclusive).
2. Receiving methadone maintenance treatment for opioid dependence at a stable once-daily dose of 80-120 mg for at least 4 weeks prior to check-in for the Inpatient Treatment Visit.
3. Body mass index ≥ 18 and ≤ 35 (kg/m2).
4. Normal screening results or abnormal results that have been deemed by the Investigator as clinically insignificant.
5. Able to understand and willing to sign an informed consent form (ICF).
6. Females practicing adequate birth control or non-childbearing potential. Medically acceptable birth control methods for this study include intrauterine device (IUD); vasectomized partner (minimum of 6 months); post-menopausal (at least 2 years); surgically sterile (at least 6 months); double barrier (diaphragm with spermicide, condoms with vaginal spermicide); abstinence; implanted or intrauterine hormonal contraceptives in use for at least 6 consecutive months prior to study dosing and throughout the study duration; and oral, patch and injected hormonal contraceptives or vaginal hormonal device (ie, NuvaRing®) in use for at least 3 consecutive months prior to study dosing and throughout the study duration.

Exclusion Criteria:

1. Abnormal cardiovascular exam at screening and before randomization, including any of the following:

   * clinically significant abnormal electrocardiogram (ECG) (eg, significant first degree atrioventricular block, complete left bundle branch block [LBBB], second or third degree heart block, clinically significant arrhythmia, or QTc interval (machine read) greater than 450 msec for males and greater than 470 msec for females)*
   * heart rate < 55 bpm or symptomatic bradycardia*
   * systolic blood pressure (SBP) < 95 mmHg or symptomatic hypotension*
   * diastolic blood pressure (DBP) < 65 mmHg*
   * blood pressure (BP) > 155/95 mmHg*
   * change in orthostatic SBP, DBP, or heart rate >25% below sitting values
   * prior history of myocardial infarction (MI) or evidence of prior MI on ECG*
   * history of long QT syndrome or relative with this condition
   * history of syncopal episodes
   * intraventricular conduction delay with QRS duration >120 ms
   * evidence of ventricular pre-excitation (eg, Wolff Parkinson White syndrome) *ECGs and vitals may be repeated as appropriate in order to confirm values and rule out extraneous results.
2. History or presence of significant or clinically unstable cardiovascular (including atrial fibrillation, congestive heart failure, myocardial ischemia, indwelling pacemaker), hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, psychiatric, neurologic, or dermatologic disease.
3. History or presence of any degree of chronic obstructive pulmonary disease.
4. History of suicidal ideations or depression requiring professional intervention including counseling or antidepressant medication over the past 12 months.
5. Positive drug (urine)/alcohol (breath) test at screening or check-in excluding methadone. Subjects who have a positive test for heroin and benzodiazepines at the Screening Visit may be enrolled if the test is negative at check-in to the Inpatient Treatment Visit. Subjects who have a positive test for heroin or benzodiazepines at the Screening Visit must sign an ICF at check-in to the Inpatient Clinic Visit.
6. Receiving methadone for pain management.
7. Positive test for human immunodeficiency virus (HIV) or hepatitis B surface antigen (HBsAg). Subjects with a positive test for hepatitis C antibodies (HCV) may be enrolled if subject is asymptomatic.
8. Estimated creatinine clearance < 80 mL/minute at screening (Cockcroft-Gault formula).
9. AST, ALT, or alkaline phosphatase > 3.0 x upper limit of normal at screening or check-in.
10. Amylase or lipase > 1.5 x upper limit normal at screening or check-in.
11. Clinically significant out-of-reference range clinical chemistry values, with particular attention to potassium, magnesium, and calcium.
12. History of hypotension.
13. History of hypersensitivity or allergy to clonidine or any clonidine analogue.
14. Use of any new prescription medication within 12 days prior to check-in.
15. Use of any over-the-counter medication, including herbal products, within the 5 days prior to check-in. Up to 2 grams per day of acetaminophen is allowed at the discretion of the principal investigator or his designee.
16. Use of any drug known to affect QTc within 30 days prior to check-in (tobacco and methadone excluded).
17. Blood donation or significant blood loss within 30 days prior to check-in.
18. Plasma donation within 7 days prior to check-in.
19. Participation in another clinical trial within 30 days prior to check-in.
20. Females who are pregnant or lactating.
21. Participation in the lofexidine hydrochloride pilot protocol USWM-LX1-1005-1.
22. Any other condition or prior therapy, which, in the opinion of the Investigator, would make the subject unsuitable for this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2012-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Changes in QTc Interval | baseline and at each escalating lofexidine dosing plateau day 3 (participant time in the study will vary based on tolerability but each dose plateau will be evaluated after 3 days at any given dose level)
  The ECG analysis will be conducted by a central laboratory under blinded review. QTc intervals at baseline (methadone maintenance dose only) will be compared to a time matched profile at each increasing lofexidine dose (as tolerated by the subjects), both before and after a withdrawal response is elicited.

SECONDARY OUTCOMES:
Change from Baseline in the Short Opioid Withdrawal Scale (SOWS) | baseline and daily assessments during methadone withdrawal phases (participant time in withdrawal will vary based on lofexidine tolerability, however on average subjects will be in a methadone withdrawal phase of the study for approximately 10 days)
  SOWS Scores at Baseline (representing when a patient is on his/her normal methadone maintenance dose when withdrawal should be minimal or zero) will be compared to SOWS Scores during methadone reduction phases of the study to determine how the intervention is affecting withdrawal. Smaller changes from baseline indicate better control of withdrawal symptoms.
Change from Baseline in the Clinical Opiate Withdrawal Scale (COWS) | baseline and daily assessments during methadone withdrawal phases (participant time in withdrawal will vary based on lofexidine tolerability, however on average subjects will be in a methadone withdrawal phase of the study for approximately 10 days)
  COWS Scores at Baseline (representing when a patient is on his/her normal methadone maintenance dose when withdrawal should be minimal or zero) will be compared to COWS Scores during methadone reduction phases of the study to determine how the intervention is affecting withdrawal. Smaller changes from baseline indicate better control of withdrawal symptoms.
Methadone Area Under the Curve (AUC) | Baseline pre-dose, 2, 3, 4, 5, 6, 10 and 24 hours; plateau days pre-dose, 0.5, 1 , 2, 3, 4, and 5 hours post dose
  AUC will be calculated for methadone at baseline and at each escalating lofexidine dosing plateau day 3 (participant time in the study will vary based on tolerability but each dose plateau will be evaluated after 3 days at any given dose level)
Lofexidine Area Under the Curve (AUC) | plateau days pre-dose, 0.5, 1 , 2, 3, 4, and 5 hours post dose
  AUC will be calculated for lofexidine at each escalating lofexidine dosing plateau day 3 (participant time in the study will vary based on tolerability but each dose plateau will be evaluated after 3 days at any given dose level)
Change in Vital Signs | baseline & 15 min prior to each dose & 3.5 hr after 8 AM, 1 and 6 PM doses on each day lofexidine dose is escalated [time in study will vary, but participants will be exposed to up 3 different lofexidine doses (from 0.4 QID to 0.8 mg QID)]
  Vital signs of subjects on methadone alone (baseline) will be compared to participant vital signs while taking methadone and the range of studied lofexidine doses.
Change in Adverse Events | baseline and during treatment visit [participant time in the study will vary, however participants will be exposed to up 3 different lofexidine doses (escalating from 0.4 QID to 0.8 mg QID) over inpatient period of up to 21 days]
  Adverse Events in subjects on methadone alone (baseline) will be compared to participant adverse events while taking methadone and the range of studied lofexidine doses.

CONTACTS AND LOCATIONS:
Overall Officials: Charles W. Gorodetzky, MD, PhD, Study Director — US WorldMeds; James A Longstreth, PhD, Study Director — US WorldMeds
Locations (1):
- Lifetree Clinical Research, Salt Lake City, Utah, United States